CLINICAL TRIAL: NCT03440372
Title: Induction Study #1 - A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Oral Ozanimod as Induction Therapy for Moderately to Severely Active Crohn's Disease
Brief Title: Induction Study #1 of Oral Ozanimod as Induction Therapy for Moderately to Severely Active Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-3201; U1111-1203-7225 (Registry Identifier: WHO); 2017-004292-31 (EudraCT Number)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Crohn Disease; Oral; Ozanimod; Moderately active; Severely active; RPC01; RPC01-3201
MeSH Terms: conditions — Crohn Disease | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Administration of oral Ozanimod (Experimental)
  Interventions: Drug: Ozanimod
- Administration of Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Arms: Administration of oral Ozanimod
Other: Placebo — Specified dose on specified days
  Arms: Administration of Placebo

SUMMARY:
This is a study to explore the effect of oral ozanimod as an induction treatment for participants with moderately to severely active Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease for ≥ 3 months on endoscopy and on histological exam
* Inadequate response or loss of response to corticosteroids, immunomodulators, and/or biologic therapies
* Crohn's Disease Activity Index (CDAI) score ≥ 220 and ≤ 450
* An average daily stool frequency ≥ 4 points and/or an abdominal pain of ≥ 2 points
* Has Simple Endoscopic Score for Crohn's Disease (SES-CD) score of ≥ 6 (or SES-CD ≥ 4 in participants with isolated ileal disease)

Exclusion Criteria:

* Has a diagnosis of ulcerative colitis, indeterminate colitis, radiation colitis, or ischemic colitis, or has strictures with prestenotic dilatation requiring procedural intervention
* Has extensive small bowel resection (>100cm) or known diagnosis of short bowel syndrome, or requires total parenteral nutrition
* Current stoma, ileal-anal pouch anastomosis, or fistula

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (408):
- United States (107):
  - Holland Center for Family Health, Peoria, Arizona
  - Local Institution - 026, North Little Rock, Arkansas
  - Local Institution - 284, Camarillo, California
  - Local Institution - 165, Chula Vista, California
  - Local Institution - 039, Garden Grove, California
  - San Diego Clinical Trials, La Mesa, California
  - Local Institution - 061, Los Angeles, California
  - Local Institution - 110, Los Angeles, California
  - Local Institution - 140, Mission Viejo, California
  - Alliance Clinical Research, Oceanside, California
  - Local Institution - 027, Orange, California
  - Palo Alto Center-Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Local Institution - 006, Rialto, California
  - Local Institution - 003, San Diego, California
  - Local Institution - 297, Lakewood, Colorado
  - Local Institution - 225, Bristol, Connecticut
  - Local Institution - 091, New Haven, Connecticut
  - Local Institution - 062, Clearwater, Florida
  - Local Institution - 218, Gainesville, Florida
  - Local Institution - 203, Hialeah, Florida
  - Harmony Medical Research Institute, Hialeah, Florida
  - Local Institution - 078, Hialeah, Florida
  - Local Institution - 179, Hollywood, Florida
  - Local Institution - 101, Homestead, Florida
  - Local Institution - 016, Largo, Florida
  - Local Institution - 199, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Local Institution - 169, Miami, Florida
  - Local Institution - 090, Naples, Florida
  - Local Institution - 214, New Smyrna Beach, Florida
  - Local Institution - 076, Orlando, Florida
  - Local Institution - 098, Port Orange, Florida
  - Local Institution - 226, Tampa, Florida
  - Local Institution - 149, Tampa, Florida
  - Local Institution - 114, Weeki Wachee, Florida
  - Local Institution - 205, Atlanta, Georgia
  - Local Institution - 222, Atlanta, Georgia
  - Local Institution - 019, Atlanta, Georgia
  - Local Institution - 063, Atlanta, Georgia
  - Local Institution - 074, Columbus, Georgia
  - Local Institution - 028, Macon, Georgia
  - Local Institution - 194, Chicago, Illinois
  - Local Institution - 036, Chicago, Illinois
  - Local Institution - 146, Urbana, Illinois
  - Iowa Digestive Disease Center, Clive, Iowa
  - Local Institution - 155, Lexington, Kentucky
  - CroNOLA LLC, Houma, Louisiana
  - Local Institution - 053, Lake Charles, Louisiana
  - Local Institution - 104, New Orleans, Louisiana
  - Local Institution - 278, Baltimore, Maryland
  - Local Institution - 129, Catonsville, Maryland
  - Local Institution - 282, Glen Burnie, Maryland
  - Local Institution - 142, Chestnut Hill, Massachusetts
  - Local Institution - 228, North Worcester, Massachusetts
  - Local Institution - 286, Springfield, Massachusetts
  - Local Institution - 191, Caro, Michigan
  - Local Institution - 108, Southfield, Michigan
  - Local Institution - 301, Wyoming, Michigan
  - Local Institution - 300, Ypsilanti, Michigan
  - Local Institution - 274, Jackson, Mississippi
  - Local Institution - 029, St Louis, Missouri
  - Local Institution - 215, Englewood, New Jersey
  - Local Institution - 144, Brooklyn, New York
  - Local Institution - 009, Great Neck, New York
  - Local Institution - 105, New York, New York
  - Local Institution - 043, New York, New York
  - Local Institution - 094, Orchard Park, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Local Institution - 017, Asheville, North Carolina
  - Local Institution - 152, Charlotte, North Carolina
  - Local Institution - 055, Charlotte, North Carolina
  - Local Institution - 133, Greenville, North Carolina
  - Local Institution - 302, Raleigh, North Carolina
  - Local Institution - 210, Beachwood, Ohio
  - Local Institution - 291, Cincinnati, Ohio
  - Local Institution - 018, Cleveland, Ohio
  - Local Institution - 177, Mentor, Ohio
  - Local Institution - 211, Warren, Ohio
  - Local Institution - 208, Oklahoma City, Oklahoma
  - Local Institution - 131, Oklahoma City, Oklahoma
  - Local Institution - 113, Portland, Oregon
  - Local Institution - 197, Hershey, Pennsylvania
  - Penn State University Milton S Hershey Medical Center, State College, Pennsylvania
  - Local Institution - 253, Providence, Rhode Island
  - Local Institution - 289, Charleston, South Carolina
  - Local Institution - 121, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - Local Institution - 158, Austin, Texas
  - Local Institution - 056, Houston, Texas
  - Local Institution - 150, Houston, Texas
  - Local Institution - 102, Houston, Texas
  - Local Institution - 082, Houston, Texas
  - Local Institution - 303, Houston, Texas
  - Local Institution - 088, Houston, Texas
  - Local Institution - 085, San Antonio, Texas
  - Local Institution - 223, San Antonio, Texas
  - Local Institution - 007, Southlake, Texas
  - Local Institution - 073, Tyler, Texas
  - Local Institution - 025, Salt Lake City, Utah
  - Local Institution - 189, Gainesville, Virginia
  - Local Institution - 298, Manassas, Virginia
  - Local Institution - 139, Petersburg, Virginia
  - Virginia Gastroenterology Institute PC, Suffolk, Virginia
  - Local Institution - 296, Williamsburg, Virginia
  - Local Institution - 125, Spokane, Washington
  - Aurora Health Care Aurora Research, Grafton, Wisconsin
- Argentina (11):
  - Local Institution - 501, Buenos Aires
  - Local Institution - 494, Buenos Aires
  - Local Institution - 571, Buenos Aires
  - Local Institution - 500, Buenos Aires
  - Local Institution - 570, Córdoba
  - Local Institution - 495, Córdoba
  - Local Institution - 569, Mar del Plata
  - Local Institution - 496, Rosario
  - Local Institution - 497, Rosario
  - Local Institution - 502, Rosario, Santa Fe
  - Local Institution - 492, San Miguel de Tucumán
- Australia (13):
  - Local Institution - 310, Concord, New South Wales
  - Local Institution - 319, Kingswood, New South Wales
  - Local Institution - 323, Wollongong, New South Wales
  - Local Institution - 707, Maroochydore, Queensland
  - Local Institution - 311, Woolloongabba, Queensland
  - Local Institution - 308, Adelaide, South Australia
  - Local Institution - 708, Adelaide, South Australia
  - Local Institution - 320, Woodville South, South Australia
  - Local Institution - 709, Melbourne, Victoria
  - Local Institution - 316, Murdoch, Western Australia
  - Local Institution - 325, Bankstown
  - Local Institution - 330, Box Hill
  - Local Institution - 324, Sydney, NSW
- Belarus (2):
  - Local Institution - 745, Grodno
  - Local Institution - 737, Vitebsk
- Belgium (8):
  - Local Institution - 943, Brasschaat, Antwerpen
  - Local Institution - 940, Brussels
  - Local Institution - 939, Edegem
  - Local Institution - 937, Ghent
  - Local Institution - 942, Leuven
  - Local Institution - 936, Liège
  - Local Institution - 938, Seraing
  - Local Institution - 941, Tournai
- Bosnia and Herzegovina (4):
  - Local Institution - 743, Banja Luka
  - Local Institution - 741, Mostar
  - Local Institution - 738, Sarajevo
  - Local Institution - 742, Sarajevo
- Bulgaria (8):
  - Local Institution - 456, Blagoevgrad
  - Local Institution - 746, Plovdiv
  - Local Institution - 747, Sofia
  - Local Institution - 627, Sofia
  - Local Institution - 749, Sofia
  - Local Institution - 748, Sofia
  - Local Institution - 553, Stara Zagora
  - Local Institution - 754, Varna
- Canada (10):
  - Local Institution - 273, Calgary, Alberta
  - Local Institution - 227, Edmonton, Alberta
  - Local Institution - 263, Kelowna, British Columbia
  - Local Institution - 255, Vancouver, British Columbia
  - Local Institution - 261, Winnipeg, Manitoba
  - Local Institution - 268, Bridgewater, Nova Scotia
  - Local Institution - 252, London, Ontario
  - Local Institution - 251, London, Ontario
  - Local Institution - 275, Toronto, Ontario
  - Local Institution - 271, Vaughan, Ontario
- Chile (5):
  - Local Institution - 389, Concepción
  - Local Institution - 392, Santiago
  - Local Institution - 387, Santiago
  - Local Institution - 391, Santiago
  - Local Institution - 390, Santiago
- Croatia (8):
  - Local Institution - 453, Koprivnica
  - Local Institution - 763, Osijek
  - Local Institution - 764, Rijeka
  - Local Institution - 765, Split
  - Local Institution - 452, Zagreb
  - Local Institution - 761, Zagreb
  - Local Institution - 762, Zagreb
  - Local Institution - 766, Zagreb
- Czechia (12):
  - Local Institution - 767, Brno
  - Local Institution - 772, Brno
  - Local Institution - 773, Hradec Králové
  - Local Institution - 775, Most
  - Local Institution - 771, Olomouc
  - Local Institution - 774, Pardubice
  - Local Institution - 769, Pilsen
  - Local Institution - 573, Prague
  - Local Institution - 368, Prague
  - Local Institution - 776, Prague
  - Local Institution - 768, Prague
  - Local Institution - 770, Prague
- Denmark (3):
  - Local Institution - 611, Copenhagen
  - Local Institution - 610, Holbæk
  - Local Institution - 609, Nykøbing Falster
- Local Institution - 614, Turku, Finland
- France (10):
  - Local Institution - 638, Amiens
  - Local Institution - 711, Créteil
  - Local Institution - 616, Dijon
  - Local Institution - 615, Grenoble
  - Local Institution - 633, Lillie Cedex
  - Local Institution - 646, Marseille
  - Local Institution - 507, Montpellier
  - Local Institution - 641, Rennes
  - Local Institution - 612, Rouen
  - Local Institution - 643, Toulouse
- Georgia (3):
  - Local Institution - 248, Tbilisi
  - Local Institution - 247, Tbilisi
  - Local Institution - 249, Tbilisi
- Germany (12):
  - Local Institution - 626, Berlin
  - Local Institution - 665, Berlin
  - Local Institution - 650, Berlin
  - Local Institution - 662, Frankfurt
  - Local Institution - 654, Frankfurt
  - Local Institution - 659, Hamburg
  - Local Institution - 651, Leipzig
  - Local Institution - 655, Ludwigshafen am Rhein
  - Local Institution - 730, Ludwigshafen am Rhein
  - Local Institution - 661, Stuttgart
  - Local Institution - 666, Tübingen
  - Local Institution - 663, Ulm
- India (11):
  - Local Institution - 444, Hyderabad, Andhra Pradesh
  - Local Institution - 407, Surat, Gujarat
  - Local Institution - 332, Gurgaon, Haryana
  - Local Institution - 445, Kochi, Kerala
  - Local Institution - 446, Ludhiana, Punjab
  - Local Institution - 443, Jaipur, Rajasthan
  - Local Institution - 399, Jaipur, Rajasthan
  - Local Institution - 408, Coimbatore, Tamil Nadu
  - Local Institution - 331, Hyderabad, Telangana
  - Local Institution - 457, Delhi
  - Local Institution - 411, New Delhi
- Ireland (2):
  - Local Institution - 975, Dublin, Dublin
  - Local Institution - 973, Dublin
- Israel (5):
  - Local Institution - 345, Bat Yam
  - Local Institution - 339, Jerusalem
  - Local Institution - 344, Nahariya
  - Local Institution - 342, Ramat Gan
  - Local Institution - 338, Rehovot
- Italy (20):
  - Local Institution - 677, Bologna
  - Local Institution - 684, Brescia
  - Local Institution - 688, Brescia
  - Local Institution - 689, Castellana Grotte
  - Local Institution - 679, Catanzaro
  - Local Institution - 687, Chieti
  - Local Institution - 674, Messina
  - Local Institution - 672, Milan
  - Local Institution - 686, Milan
  - Local Institution - 334, Milan
  - Local Institution - 678, Monza
  - Local Institution - 685, Padua
  - Local Institution - 682, Palermo
  - Local Institution - 673, Pavia
  - Local Institution - 681, Roma
  - Local Institution - 675, Roma
  - Local Institution - 671, Rome
  - Local Institution - 680, Udine
  - Local Institution - 670, Varese
  - Local Institution - 676, Verona
- Latvia (3):
  - Local Institution - 602, Riga
  - Local Institution - 601, Riga
  - Local Institution - 600, Riga
- Mexico (10):
  - Local Institution - 526, Zapapan, Jalisco
  - Local Institution - 532, Monterrey, Nuevo León
  - Local Institution - 525, Monterrey, Nuevo León
  - Local Institution - 447, Monterrey, Nuevo León
  - Local Institution - 449, Monterrey, Nuevo León
  - Local Institution - 529, Querétaro City, Querétaro
  - Local Institution - 528, Chihuahua City
  - Local Institution - 448, Mexico City
  - Local Institution - 527, México
  - Local Institution - 530, Tlalpan
- Moldova (5):
  - Local Institution - 811, Chisinau
  - Local Institution - 810, Chisinau
  - Local Institution - 809, Chisinau
  - Local Institution - 812, Chisinau
  - Local Institution - 813, Chisinau
- Poland (29):
  - Local Institution - 403, Zamość, Lublin Voivodeship
  - Local Institution - 597, Zamość, Lublin Voivodeship
  - Local Institution - 820, Bialystok
  - Local Institution - 818, Bochnia
  - Local Institution - 238, Katowice
  - Local Institution - 828, Katowice
  - Local Institution - 819, Katowice
  - Local Institution - 815, Krakow
  - Local Institution - 823, Krakow
  - Local Institution - 826, Krakow
  - Local Institution - 817, Kłodzko
  - Local Institution - 829, Lodz
  - Local Institution - 888, Lodz
  - Local Institution - 760, Lublin
  - Local Institution - 830, Olsztyn
  - Local Institution - 402, Opole
  - Local Institution - 400, Oświęcim
  - Local Institution - 758, Poznan
  - Local Institution - 575, Poznan
  - Local Institution - 401, Poznan
  - Local Institution - 239, Sopot
  - Local Institution - 235, Szczecin
  - Local Institution - 822, Torun
  - Local Institution - 824, Tychy
  - Local Institution - 827, Ul. Piotrkowska 177
  - Local Institution - 410, Warsaw
  - Local Institution - 576, Warsaw
  - Local Institution - 825, Warsaw
  - Local Institution - 236, Warsaw
- Romania (10):
  - Local Institution - 808, Bucharest
  - Local Institution - 836, Bucharest
  - Local Institution - 499, Bucharest
  - Local Institution - 795, Bucharest
  - Local Institution - 837, Bucharest
  - Local Institution - 839, Bucharest
  - Local Institution - 842, Bucharest
  - Local Institution - 838, Cluj-Napoca
  - Local Institution - 843, Craiova
  - Local Institution - 840, Târgu Mureş
- Russia (24):
  - Local Institution - 598, Chita
  - Local Institution - 848, Irkutsk
  - Local Institution - 892, Kazan'
  - Local Institution - 599, Khanty-Mansiysk
  - Local Institution - 927, Krasnoyarsk
  - Local Institution - 851, Moscow
  - Local Institution - 594, Novosibirsk
  - Local Institution - 858, Petrozavodsk
  - Local Institution - 859, Pushkin
  - Local Institution - 960, Pyatigorsk
  - Local Institution - 846, Pyatigorsk
  - Local Institution - 883, Rostov-on-Don
  - Local Institution - 862, Saint Petersburg
  - Local Institution - 847, Saint Petersburg
  - Local Institution - 857, Saint Petersburg
  - Local Institution - 845, Saint Petersburg
  - Local Institution - 856, Saint Petersburg
  - Local Institution - 844, Samara
  - Local Institution - 806, Tula
  - Local Institution - 861, Ufa
  - Local Institution - 855, Veliky Novgorod
  - Local Institution - 935, Vladimir
  - Local Institution - 999, Vladivostok
  - Local Institution - 986, Vladivostok
- Saudi Arabia (4):
  - Local Institution - 534, Dammam
  - Local Institution - 537, Jeddah
  - Local Institution - 536, Riyadh
  - Local Institution - 535, Riyadh
- Serbia (3):
  - Local Institution - 241, Belgrade
  - Local Institution - 245, Belgrade
  - Local Institution - 246, Belgrade
- South Korea (10):
  - Local Institution - 437, Ansan
  - Local Institution - 441, Busan
  - Local Institution - 435, Guri-si
  - Local Institution - 436, Seongnam-si
  - Local Institution - 433, Seoul
  - Local Institution - 440, Seoul
  - Local Institution - 430, Seoul
  - Local Institution - 442, Seoul
  - Local Institution - 427, Seoul
  - Local Institution - 439, Seoul
- Spain (8):
  - Local Institution - 703, Alicante
  - Local Institution - 690, Badalona
  - Local Institution - 691, Madrid
  - Local Institution - 692, Madrid
  - Local Institution - 698, San Cristóbal de La Laguna
  - Local Institution - 696, Seville
  - Local Institution - 705, Seville
  - Local Institution - 700, Viladecans
- Switzerland (3):
  - Local Institution - 967, Bern
  - Local Institution - 968, Sankt Gallen
  - Local Institution - 969, Zurich
- Local Institution - 363, Kozlu, Taiwan
- Turkey (Türkiye) (6):
  - Local Institution - 356, Ankara
  - Local Institution - 360, Bursa
  - Local Institution - 362, Istanbul
  - Local Institution - 355, Istanbul
  - Local Institution - 354, Izmit/Kocaeli
  - Local Institution - 359, Trabzon
- Ukraine (22):
  - Local Institution - 914, Chernivtsi
  - Local Institution - 950, Dnipropetrovsk
  - Local Institution - 229, Ivano-Frankivsk
  - Local Institution - 912, Ivano-Frankivsk
  - Local Institution - 919, Kharkiv
  - Local Institution - 901, Kyiv
  - Local Institution - 915, Kyiv
  - Local Institution - 243, Kyiv
  - Local Institution - 911, Kyiv
  - Local Institution - 244, Kyiv
  - Local Institution - 918, Kyiv
  - Local Institution - 908, Kyiv
  - Local Institution - 562, Kyiv
  - Local Institution - 240, Lutsk
  - Local Institution - 234, Lviv
  - Local Institution - 910, Lviv
  - Local Institution - 242, Odesa
  - Local Institution - 905, Poltava
  - Local Institution - 934, Ternopil
  - Local Institution - 909, Vinnytsia
  - Local Institution - 224, Vinnytsia
  - Local Institution - 971, Vinnytsia
- United Kingdom (15):
  - Local Institution - 723, Southampton, Hampshire
  - Local Institution - 729, London, LND
  - Local Institution - 557, Birmingham
  - Local Institution - 714, Bristol
  - Local Institution - 560, Cardiff
  - Local Institution - 558, Chorley
  - Local Institution - 559, Corbridge Road
  - Local Institution - 712, Dundonald
  - Local Institution - 713, Glasgow
  - Local Institution - 716, Lancashire Blackpool
  - Local Institution - 722, London
  - Local Institution - 715, London
  - Local Institution - 561, North Manchester Science Park
  - Local Institution - 593, Shrewsbury
  - Local Institution - 718, Torquay

REFERENCES:
- [Derived] Feagan BG, Schreiber S, Afzali A, Rieder F, Hyams J, Kollengode K, Pearlman J, Son V, Marta C, Wolf DC, D'Haens GG. Ozanimod as a novel oral small molecule therapy for the treatment of Crohn's disease: The YELLOWSTONE clinical trial program. Contemp Clin Trials. 2022 Nov;122:106958. doi: 10.1016/j.cct.2022.106958. Epub 2022 Oct 5. PMID 36208720
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 625 participants were randomized and of these 623 received at least one dose of study treatment.
Groups:
- Treatment 1: Participants received ozanimod 0.92 mg
- Treatment 2: Participants received ozanimod matching placebo
Period: Pre-Treatment
Arm/Group | Treatment 1 | Treatment 2
Started (Started = Randomized) | 417 | 208
Completed (Completed = Treated) | 416 | 207
Not Completed | 1 | 1
Period: Treatment
Arm/Group | Treatment 1 | Treatment 2
Started (Started = Treated) | 416 | 207
Completed | 378 | 185
Not Completed | 38 | 22
Not completed — Adverse Event | 16 | 8
Not completed — Lack of Efficacy | 4 | 2
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Study Terminated by Sponsor | 2 | 1
Not completed — Other Reason | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 417 | 208 | 625
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 394 | 199 | 593
  >=65 years | 23 | 9 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 97 | 307
  Male | 207 | 111 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 34
  Not Hispanic or Latino | 391 | 190 | 581
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 21 | 9 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 378 | 188 | 566
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Crohn's Disease Activity Index (CDAI) Score < 150 at Week 12
Description: Crohn's Disease Activity Index (CDAI) is a composite score used to measure the clinical activity of Crohn's disease. CDAI uses 8 variables: number of soft/liquid stools, severity of abdominal pain (0=none to 3=severe), general well-being (0=well to 4=terrible), presence of complications, need for antidiarrheal drugs, presence of abdominal mass, hematocrit, and change in body weight. Scores for stool number, abdominal pain, and well-being are summed over the 7 days before each visit. The other factors are also recorded and weighted to create a total CDAI score, which ranges from 0-600, with higher scores indicating worse disease (score 150-219 = mild, 220-450 = moderate, >450 = severe). This measure reports the percentage of participants whose CDAI score was below 150 at 12 weeks.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 31.3 | 20.8
  Non-Responders | 64.4 | 73.4
  Imputed Non-Responders | 4.3 | 5.8
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0049, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.19 to 2.70]

2. Secondary Outcome: Percent of Participants With Average Daily Abdominal Pain Score ≤ 1 Point, and Average Daily Stool Frequency Score ≤ 3 Points With Abdominal Pain and Stool Frequency no Worse Than Baseline at Week 12
Description: Abdominal pain (AP) and stool frequency (SF) clinical remission was defined as an average daily abdominal pain score ≤1 and average daily stool frequency ≤3, with AP and SF no worse than baseline at Week 12. AP was graded on a scale from 0 (none) to 3 (severe), and SF was defined as the number of liquid or soft stools per day. This measure reports the percentage of participants who, by Week 12, had low abdominal pain (score ≤1) and three or fewer bowel movements per day, without worsening symptoms compared to when they started the study. Participants began using the diary at the first visit and continued throughout the study.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 30.5 | 21.7
  Non-Responders | 66.3 | 72.5
  Imputed Non-Responders | 3.1 | 5.8
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0179, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.09 to 2.43]

3. Secondary Outcome: Percent of Participants With a Simple Endoscopic Score for Crohn's Disease (SES-CD) Score Decrease From Baseline of ≥ 50% at Week 12
Description: The Simple Endoscopic Score for Crohn's Disease (SES-CD) is used to assess the degree of inflammation in patients with Crohn's disease. The SES-CD evaluates four components-size of ulcers, ulcerated surface, affected surface, and presence of narrowing-each scored from 0 (none) to 3 (severe): score ranges from 0-12 across four components and 0-60 overall across five segments (ileum, right colon, transverse colon, left colon, rectum). The total higher SES-CD score indicating greater inflammation. Baseline is defined as the last assessment prior to the first drug administration (based on the time of measurement, if available; otherwise, the last assessment prior to or on the date of first drug administration). This measure reports the percentage of participants whose SES-CD score improved by 50% or more from baseline to Week 12.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 22.1 | 18.4
  Non-Responders | 71.6 | 77.3
  Imputed Non-Responders | 6.3 | 4.3
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.2720, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.83 to 1.93]

4. Secondary Outcome: Percent of Participants With Crohn's Disease Activity Index (CDAI) Reduction From Baseline of ≥ 100 Points or CDAI Score < 150 at Week 12
Description: The Crohn's Disease Activity Index (CDAI) is a composite score used to measure the clinical activity of Crohn's disease. CDAI is calculated using 8 variables: number of soft/liquid stools, severity of abdominal pain (0 [none] to 3 [severe]), general well-being (0 [well] to 4 [terrible]), presence of complications, use of antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. Scores for stool frequency, pain, and well-being are summed over the 7 days prior to each visit. The remaining variables are also weighted and included in the total CDAI score, which ranges from 0-600, with higher scores indicating worse disease activity (score 150-219 = mild, 220-450 = moderate, >450 = severe). This measure reports the percentage of participants whose CDAI score improved by at least 100 points, or was below 150, at 12 weeks.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 48.8 | 39.1
  Non-Responders | 46.9 | 55.1
  Imputed Non-Responders | 4.3 | 5.8
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0193, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.07 to 2.15]

5. Secondary Outcome: Percent of Participants With Crohn's Disease Activity Index (CDAI) Reduction From Baseline of ≥ 100 Points or CDAI Score < 150 and Simple Endoscopic Score for Crohn's Disease (SES-CD) Decrease From Baseline of ≥ 50% at Week 12
Description: The Crohn's Disease Activity Index (CDAI) is a composite score used to measure clinical activity in Crohn's disease. CDAI is based on 8 variables: number of soft/liquid stools, severity of abdominal pain (0 [none] to 3 [severe]), general well-being (0 [well] to 4 [terrible]), presence of complications, use of antidiarrheal drugs, abdominal mass, hematocrit, and deviation in body weight. Scores for stool frequency, pain, and well-being are summed over 7 days prior to each visit. The total CDAI score ranges from 0-600, with higher scores indicating worse disease activity (score 150-219 = mild, 220-450 = moderate, >450 = severe). This measure reports the percentage of participants whose Crohn's disease improved at 12 weeks, defined as a CDAI decrease of at least 100 points or a score below 150, along with at least a 50% reduction in intestinal inflammation (SES-CD score).
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 16.6 | 13.5
  Non-Responders | 78.6 | 84.1
  Imputed Non-Responders | 4.8 | 2.4
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.3167, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.79 to 2.05]

6. Secondary Outcome: Percent of Participants With Crohn's Disease Activity Index (CDAI) Score < 150 at Week 12 and Simple Endoscopic Score for Crohn's Disease (SES-CD) Decrease From Baseline of ≥ 50% at Week 12
Description: This endpoint measured the percentage of participants who achieved both clinical remission and significant endoscopic improvement at Week 12. Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score of less than 150 at Week 12. Endoscopic improvement was defined as a decrease of at least 50% from baseline in the Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12. The CDAI was a composite score assessing disease activity based on symptoms and laboratory values, while the SES-CD evaluated endoscopic findings in the intestinal mucosa. Achieving both criteria indicated substantial improvement in both symptoms and intestinal inflammation.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percent of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percent of Participants
  Responders | 16.6 | 13.5
  Non-Responders | 78.6 | 84.1
  Imputed Non-Responders | 4.8 | 2.4
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.3167, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.79 to 2.05]

7. Secondary Outcome: Percent of Participants With an Average Daily Abdominal Pain Score ≤ 1 Point, and Average Daily Stool Frequency Score ≤ 3 Points With Abdominal Pain and Stool Frequency no Worse Than Baseline and an SES-CD ≤ 4 Points and Decrease ≥ 2 Points at Week 12
Description: This measure reports the percentage of participants whose Crohn's disease symptoms and gut inflammation improved at 12 weeks. It includes those with mild or no belly pain (score ≤1), no more than three bowel movements per day (score ≤3), and no worsening from baseline. It also includes participants whose gut inflammation, measured by SES-CD, was low (score ≤4) and improved by at least 2 points. SES-CD assesses inflammation based on four components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing, each scored from 0 (none) to 3 (severe) across five segments (ileum, right colon, transverse colon, left colon, rectum). The total SES-CD score ranges from 0-12 per segment and 0-60 overall, with higher scores indicating greater inflammation.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 8.7 | 6.3
  Non-Responders | 88.0 | 91.3
  Imputed Non-Responders | 3.4 | 2.4
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.2978, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.73 to 2.77]

8. Secondary Outcome: Percent of Participants With an Average Daily Abdominal Pain Score ≤ 1 Point, and Average Daily Stool Frequency Score ≤ 3 Points With Abdominal Pain and Stool Frequency Score no Worse Than Baseline and an SES-CD Decrease From Baseline of ≥ 50% at Week 12
Description: This measure reports the percentage of participants whose Crohn's disease symptoms and gut inflammation improved at 12 weeks. It includes those with mild or no belly pain (score ≤1), no more than three bowel movements per day (score ≤3), and no worsening from baseline. It also includes participants whose gut inflammation, measured by SES-CD, improved by at least 50% from baseline. SES-CD assesses inflammation based on four components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing, each scored from 0 (none) to 3 (severe): score ranges from 0-12 across four components and 0-60 overall across five segments (ileum, right colon, transverse colon, left colon, rectum). The total higher SES-CD score indicating greater inflammation.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 11.1 | 7.7
  Non-Responders | 85.6 | 89.9
  Imputed Non-Responders | 3.4 | 2.4
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.1895, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.82 to 2.72]

9. Secondary Outcome: Histologic Improvement Based on Differences Between Ozanimod and Placebo in Histologic Disease Activity Scores (ie, Global Histologic Activity Score (GHAS) Changes) at Week 12
Description: This measure evaluated improvement in gut inflammation at 12 wks using Global Histologic Activity Score (GHAS). GHAS was assessed for each ileal & colonic segment (ileum, right colon, transverse colon, left colon-descending/sigmoid colon & rectum). Segment subscores were calculated by adding scores for epithelial damage/tissue changes(0-2), cellular infiltration for mononuclear & polymorphonuclear cells(0-2 each), presence of certain cells(0-3) & erosion, ulcers, granulomas(0 or 1). GHAS score within each segment ranged from 0-16 & across five segments ranged from 0-80. Higher scores indicated more inflammation. Responders with histologic remission was defined as GHAS score ≤8 (each segment) [meeting criteria: epithelial damage(0), architectural changes(0-2), mononuclear cell infiltration(0-2), polymorphonuclear cell infiltration(0), polymorphonuclear cells in epithelium(0), erosion/ulcers(0), granuloma(0-1) & affected biopsy specimens(0-3)] & ≤40 (across all segments).
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 14.9 | 9.2
  Non-Responders | 78.4 | 85.5
  Imputed Non-Responders | 6.7 | 5.3
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0452, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.00 to 2.97]

10. Secondary Outcome: Percent of Participants With Crohn's Disease Activity Index (CDAI) Reduction From Baseline of ≥ 70 Points at Week 12
Description: This measure reports the percentage of participants whose Crohn's disease symptoms improved meaningfully after 12 weeks of treatment, defined as a decrease of at least 70 points in their Crohn's Disease Activity Index (CDAI) score from baseline. The CDAI is a composite score used to assess clinical activity in Crohn's disease, based on 8 variables: number of soft/liquid stools, severity of abdominal pain (0 [none] to 3 [severe]), general well-being (0 [well] to 4 [terrible]), presence of complications, use of antidiarrheal drugs, presence of an abdominal mass, hematocrit, and deviation in body weight. Scores for stool frequency, pain, and well-being are summed over 7 days prior to each visit. The total CDAI score ranges from 0-600, with higher scores indicating more severe disease (score 150-219 = mild, 220-450 = moderate, >450 = severe).
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 55.3 | 45.4
  Non-Responders | 40.4 | 48.8
  Imputed Non-Responders | 4.3 | 5.8
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0173, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.08 to 2.14]

11. Secondary Outcome: Percent of Participants With Absence of Ulcers ≥ 0.5 cm With No Segment With Any Ulcerated Surface ≥ 10% at Week 12
Description: This measure shows the percentage of participants have no longer any large ulcers (bigger than 0.5 cm) in their gut and in any section of the gut, less than 10% of the surface has ulcers at 12 weeks. This helps to understand how well the treatment is healing the gut and reducing ulceration.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 26.9 | 20.3
  Non-Responders | 66.8 | 75.4
  Imputed Non-Responders | 6.3 | 4.3
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0670, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.97 to 2.20]

12. Secondary Outcome: Percent of Participants With a Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline of ≥ 50% at Week 12
Description: CDEIS is an index used to determine Crohn's disease severity by endoscopic exam of the ileum and colon. The intestine is divided into 5 segments: rectum, sigmoid/left colon, transverse colon, right colon, and ileum. In each segment, four variables are assessed: deep ulceration, superficial ulceration, percentage of ulcerated surface, and percentage of surface affected by Crohn's disease, using 10-cm visual analogue scales. The presence of ulcerated and nonulcerated stenosis is also evaluated across the entire intestine. These factors are weighted and summed for a total score from 0-44, with higher scores indicating more severe disease. This measure reports the percentage of participants whose CDEIS score improved by at least 50% at 12 weeks, based on endoscopic exam.
Time Frame: At Week 12
Population: Intent to treat population consist of all randomized participants that received at least 1 dose of investigational drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 416 | 207
Percentage of Participants
  Responders | 25.5 | 19.3
  Non-Responders | 68.3 | 76.3
  Imputed Non-Responders | 6.3 | 4.3
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority; p = 0.0835, Mantel Haenszel; Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.95 to 2.16]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality, Serious Adverse Events (SAEs) and Other Adverse Events (AEs) were assessed from first dose of study medication until study completion (assessed up to approximately 79 months).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Treatment 1 | Treatment 2
All-Cause Mortality (participants affected / at risk) | 0/416 | 0/207
Serious Adverse Events (participants affected / at risk) | 27/416 | 10/207
Other Adverse Events (participants affected / at risk) | 22/416 | 22/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=416) | Treatment 2 (N=207)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 10 | 4
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=416) | Treatment 2 (N=207)
Crohn's disease (Gastrointestinal disorders) | 9 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03440372/Prot_SAP_000.pdf